CLINICAL TRIAL: NCT00463879
Title: Galantamine for Cognitive Deficits in Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0508000458
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Smoking; Galantamine; Nicotine; Cognitive Deficits
MeSH Terms: conditions — Schizophrenia; Smoking; Cognition Disorders | interventions — Galantamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
The purpose of this study is to determine the acute effects of the nicotinic receptor allosteric modulator galantamine (0, 4 and 8 mg) on neurocognitive function in schizophrenic smokers (n=20) versus schizophrenic nonsmokers (n=10) in an outpatient human laboratory setting.

DETAILED DESCRIPTION:
The proposed study will entail a comprehensive evaluation of the effects of acute doses of the nAChR allosteric modulator galantamine hydrochloride (0, 4 and 8 mg) on neurocognitive measures in schizophrenic smokers (n=20) and schizophrenic non-smokers (n=10) in a human laboratory paradigm. After training on a battery of neurocognitive assessments, all subjects will be studied during three separate test weeks where they will complete the neurocognitive batter at baseline, and then again after acute administration of the three doses of galantamine in a counterbalanced order across subjects in each experimental group. Specifically, smokers would be randomized into one of two groups: 1) those who undergo overnight smoking abstinence prior to the study cognitive sessions in order to determine galantamine's effects on abstinence-induced cognitive impairment, and 2) those who may smoke as usual prior to the study cognitive sessions. The inclusion of nonsmokers will allow for the assessment of galantamine's effects on cognitive deficits in schizophrenia independent of cigarette smoking. Finally, genetic variations in key metabolic genes involved in catecholamine metabolism (COMT and DBH) would be evaluated as determinants of galantamine-related improvements in cognitive performance in schizophrenic smokers and nonsmokers.

We predict that galantamine will dose-dependently improve selected cognitive deficits associated with schizophrenia (e.g., spatial working memory, sustained attention and prepulse inhibition) which we have previously shown are selectively improved by cigarette smoking in smokers with schizophrenia [18], and that this effect would be more pronounced in nonsmokers with schizophrenia. If our results are positive, they would support the rationale for controlled clinical trials using nAChR agonists like galantamine to treat selected domains of cognitive dysfunction in this disorder.

Study Design:

The following experimental groups will be studied:

1. Schizophrenic Smokers under abstinence conditions (n=10)
2. Schizophrenic Smokers in the smoking condition. (n=10)
3. Schizophrenic Nonsmokers (n=10)

Three acute doses of galantamine (GAL) will be tested (0, 4 and 8 mg) in all subjects during three separate test sessions separated by at least 3 days, with study medication doses across sequential subjects given in a randomized, counterbalanced manner.

Smokers (n=20) and nonsmokers (n=10) with schizophrenia will be recruited from the outpatient division of The Connecticut Mental Health Center (CMHC) in New Haven, CT, and it's affiliated satellite centers (Hispanic Clinic, West Haven Mental Health Center, and Yale Behavioral Mental Health Center).

Screening Procedures:

All potential subjects would meet with study staff over 2-3 intake and evaluation sessions to determine study eligibility, which would typically take place within 4 weeks of study enrollment. A description of the evaluation measures is given below:

The screening evaluation will include completion of informed consent forms, a urine toxicology screen to screen for recent use of illegal substances, a urine pregnancy test for female subjects, a psychiatric evaluation using the SCID for DSM-IV disorders, PANSS, AIMS, Webster, Barnes, BDI, Tiffany Questionnaire for Smoking Urges (T-QSU), Minnesota Nicotine Withdrawal Scale (M-NWS), Shipley Full Scale Intelligence Quotient (IQ), a blood draw for plasma nicotine, plasma cotinine, as well as CBC and LFT's, and a physical examination conducted by Dr. George. Subjects will be separately consented for the genetics portion of the study and blood will be taken for genotyping purposes. Finally, a pre-study neuropsychological testing session would be performed in order to orient and train participants on the laboratory procedures. Subjects who are pregnant or planning on becoming pregnant will not be eligible to participate.

We will compensate all subjects who complete the screening and evaluation process ($25.00) and the neurocognitive training session ($25.00) for a total of $50.00. In addition, subjects would be paid $25.00 for donating a blood sample for genotyping.

Blood for genotyping will be obtained for COMT and DBH polymorphisms in smokers and nonsmokers in schizophrenia participating in this study. The genotyping for these studies will be done in collaboration with the Psychiatric Genetics laboratory of Joseph F. Cubells, M.D., Ph.D. at Emory University.

Experimental Procedures: Smokers will be tested on the cognitive battery at baseline (Day 1, with periodic smoking breaks to minimize nicotine withdrawal), and then again 24 hours later after overnight smoking abstinence (Day 2). Non-smokers will be tested at baseline (Day 1) and again 24 hours later (Day 2). Study medications will be given as a single dose before the Day 2 session which will produce ascending plasma drug levels (t= ½ 5/7 h) during the two hour testing session, in a counterbalanced dosing schedule of galantamine hydrobromide (0, 4, and 8 mg) within each test group. If systolic blood pressure is below 90 mm Hg, the galantamine study medication will be held. Before and after each session (Day 1 and Day 2), clinical ratings using the PANSS, HDRS, extrapyramidal ratings, and adverse event ratings would be completed. For smokers, pre-session tobacco craving and withdrawal ratings, expired breath carbon monoxide, and plasma cotinine and nicotine levels would be obtained. Smokers randomized to the abstinence condition would receive $150.00 for successful completion of each of the subsequent three test session procedures requiring overnight abstinence ($50.00 for successful abstinence, and $100.00 for subsequent testing session completion). Smokers randomized to the non-abstinence condition would be also receiving $150.00 for successful completion of each of the three test session procedures in order to maintain consistency. Nonsmokers would receive $100.00 for completion of each of the three test sessions beyond the training session. In addition, a completion bonus of $50.00 will be paid to all subjects who complete all study procedures. Thus, smokers with schizophrenia could earn $575.00, and nonsmokers $425.00 for their completion of the entire study. The proposed single subject timeline is given below:

ELIGIBILITY:
Inclusion Criteria:

-

Schizophrenic smokers (n=20) and schizophrenic nonsmokers (n=10) in these studies (total n=20 subjects) will be:

1. Between 18 and 60 years of age,
2. Have a Full Scale IQ score >80.
3. Smokers will meet DSM-IV criteria for nicotine dependence, and smoke at least 15 cigarettes per day, with an FTND score at baseline >5, breath CO >10, and plasma cotinine >150 ng/ml.
4. Nonsmokers will report a history of never smoking (<100 cigarettes lifetime) or be abstinent from smoking for at least 6 months prior to randomization, with abstinence biochemically confirmed by CO level <10 ppm and plasma cotinine <15 ng/ml.
5. Schizophrenic subjects will meet DSM-IV criteria for schizophrenia or schizoaffective disorder, and be on a stable dose of antipsychotic medication for at least three months, with positive symptoms stability as judged by the investigator.
6. Subjects must be non-treatment seeking smokers with respect to their nicotine dependence.

Exclusion Criteria:

1. Meet criteria for current abuse or dependence for any other alcohol or substance of abuse within the past 6 months, with the exception of nicotine dependence (smokers) or caffeine (all groups).
2. An inability to learn the neuropsychological tasks during the training session.
3. History of dementia, other neurological illness (e.g. idiopathic Parkinson's Disease, Epilepsy), or any other acute or chronic medical condition known to significantly influence neurocognitive function, at the discretion of the P.I. and Project Director.
4. A history of severe renal or hepatic insufficiency, or a known hypersensitivity to galantamine hydrochloride (Razadyne®).
5. For smokers, current use of any tobacco products (chewing tobacco, cigars, nicotine replacement therapies like lozenges, gum, nasal spray, inhaler or patch) besides cigarettes.
6. A history of hypotension, or currently taking anti-hypertensive medication.
7. Interested in quitting smoking (in which case they will be referred to our smoking cessation treatment study).
8. Not capable of giving informed consent for participation in this study.
9. Positive urine toxicology screen for any substance of abuse.
10. Patients who are pregnant or planning on becoming pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
1. Change on selected cognitive deficits associated with schizophrenia (e.g., spatial working memory, sustained attention and prepulse inhibition.)

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D., Principal Investigator — University of Toronto
Locations (1):
- Connecticut Mental Health Center, Yale School of Medicine, New Haven, Connecticut, United States